CLINICAL TRIAL: NCT02454582
Title: Effect of Non-invasive Ventilation (NIV) on Cerebral Oxygenation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ass.-Prof. PD Dr. Klaus Ulrich Klein (Other)
Responsible Party: Sponsor-Investigator, Ass.-Prof. PD Dr. Klaus Ulrich Klein, Ass.-Prof. PD Dr. Klaus Ulrich Klein, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: EK Number: 1264/2014
Record Dates: First submitted 2015-05-19; First posted 2015-05-27 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Insufficiency
MeSH Terms: conditions — Respiratory Insufficiency

ARMS (2):
- Group 1 (Other): 15min without CPAP, then 15min with CPAP NIRS measurement, Somanetics INVOS Cerebral Oxymeter 5100C
  Interventions: Device: Somanetics INVOS Cerebral Oxymeter 5100C
- Group 2 (Other): 15min with CPAP, then 15min without CPAP NIRS measurement, Somanetics INVOS Cerebral Oxymeter 5100C
  Interventions: Device: Somanetics INVOS Cerebral Oxymeter 5100C

INTERVENTIONS:
Device: Somanetics INVOS Cerebral Oxymeter 5100C — Non- invasive transcranial near infrared cerebral oxygenation with or without CPAP

SUMMARY:
SUMMARY AND AIM

Background:

The proper management of brain oxygenation is an essential component of all anaesthesiologic procedures. Nevertheless, the brain remains one of the least monitored organs in the perioperative phase and intensive care therapy.

The INVOS Brain Oxymeter (IBO) is a reliable trend monitor for changes in regional cerebral oxygenation (rSO2).

It is a current assumption that rSO2 directly correlates with Sa02, which can be influenced by different ventilation assistance systems, e.g. CPAP therapy.

Objectives:

The project aims at investigating changes of rSO2 in patients undergoing CPAP therapy for max. 15 minutes, in order to evaluate the effect of CPAP on cerebral oxygenation.

Methods:

NIRS measurement (with IBO) will be performed on the temporoparietal cortex on both sides of the head. The trial will consist of two parts i.e. with or without ventilatory assistance. The order of starting the study with or without CPAP therapy will be randomized. During each part the measurements will be performed until reaching a steady state (no change in rSO2 ± 2% for 3 min) but with a maximum duration of 15min. After each interval a BGA (blood gas analysis) will be performed.

DETAILED DESCRIPTION:
BACKGROUND

Near infrared spectroscopy (NIRS) is a non-invasive method for the measurement of blood flow in tissues, first used for cerebral tissue oxygenation in 1977. 1 NIRS is a spectroscopic technique, which uses electromagnetic waves (700-950nm), an emitter and a detector. In the last 20 years there was an enormous development in the instrumentation and application of NIRS. This technique now allows for measuring the oxygenation of the brain tissue. 2-13 The INVOS Brain Oxymeter (IBO) is a reliable trend monitor for changes in regional cerebral oxygenation (rSO2) and correlates with the hemoglobin saturation in venous, capillary and arterial blood, using an algorithm based upon the Beer-Lambert law. 4,14 The IBO system uses light, with wavelengths between 730-810 nm, that penetrates layers of the human body, among them the skin, the scull and the brain. It is either scattered within the tissue or absorbed by present chromophores. In the rather transparent near infrared region, there are many absorbing light chromophores, but only three are important as far as the oxygenation is concerned, namely hemoglobin (HbO2), deoxyhemoglobin (Hb) and cytochrome oxidase (CtOx). Oxygenated and deoxygenated hemoglobin absorb light at different wavelengths, allowing a differentiation of these two forms of hemoglobin.15 The sensors, ("SomaSensors"), are applied to the patient's forehead with an integrated medical-grade adhesive.16 The method is applied by using two source-detector distances in the sensor: a "near" one (shallow), 3 cm from the source and a "far" one (deep), 4 cm from the source. Both samples penetrate the tissue beneath the light source equally well, with the difference that the 4cm source-detector measures signals deeper in the brain.8,17 The subtraction of the near sample from the far one should leave a signal originating predominantly from the brain cortex. 16 The proper management of brain oxygenation is an essential component of all anaesthesiologic procedures. Nevertheless, the brain remains one of the least monitored organs during the perioperative phase and intensive care therapy. Up until now, the anaesthesiological application of NIRS as a method for measuring the cerebral oxygenation has only been investigated in patients undergoing cardiac surgery or cerebrovascular surgery, elderly patients undergoing major abdominal surgery and neonatal infants. 18-21 These studies indicate that the measured cerebral oxygenation is affected by the relative proportion of blood in the arterial or venous part of the capillary bed, the hemoglobin concentration and the systemic saturation in addition to the cardiac output. The precise consequences of alterations in the systemic saturation (SaO2) on the cerebral oxygenation (rSO2) remain unknown. It is a current assumption that rSO2 is directly associated with Sa02, so that an increase of SaO2 also leads to an increase of rSO2. The amount of oxygen in the arterial blood depends on the inspired oxygen and the pulmonary gas exchange. These two parameters are primarily affected by the individual's respiratory ventilation. Patients with chronic respiratory failure, or just a temporary (acute) breathing deficiency (e.g. after general anesthesia), are routinely treated with continuous positive airway pressure (CPAP) therapy. It is also commonly used in the treatment of sleep apnea and in neonates (especially premature infants). In these patients CPAP ventilation may prevent the need of tracheal (re-) intubation, or enable earlier extubation.

CPAP therapy was developed by Dr. George Gregory and colleagues in the neonatal ICU at the University of California, San Francisco in 1971 22, and then modified by Professor Colin Sullivan at Royal Prince Alfred Hospital in Sydney, Australia, in 1981. 23 Initially the CPAP therapy was mainly used for the treatment of obstructive sleep apnea at home. Nowadays it is commonly applied in ICUs as a form of non-invasive mechanical ventilation. There it is usually reserved for subgroups of patients where the oxygen treatment via a facemask is insufficient. Patients on CPAP therapy are closely monitored in the ICU setting. The treatment supports the patient's spontaneous breathing by building up a positive end expiratory pressure (PEEP). The pressure required by most patients ranges between 5 and 12 cmH2O. The patient can individually determine his or her own respiratory frequency as well as the depth of respiration.

Objectives:

The primary study goal is the investigation of the effect of CPAP therapy on rSO2 in relation to the vital parameters, hemoglobin, SaO2 (analyzed by BGA) and SpO2. These combined measurements can be used to further describe the effect of CPAP therapy on rSO2. So far, this kind of study has not been performed on patients in the ICU. Therefore, this project aims at gaining new insights into the influence of CPAP therapy on the cerebral saturation. Additionally, differences in SaO2 and vital parameters will be correlated to the rSO2. Also the occurrence of vomiting and nausea, headache and agitation during the CPAP therapy will be registered.

The following parameters will be measured, calculated and noted in the CRF (case report form):

* Blood pressure (BP)
* Heart rate (HR) and rhythm
* rSO2 (left and right hemisphere)
* BGA: arterial partial pressure of oxygen (PaO2)
* BGA: pH, Electrolytes (Na, K, Ca), Glucose, Lactate, SaO2
* BGA: Hb, Hk, MetHb, CoHb, SO2, pCO2, BE, SBC
* Ventilation: CPAP, MV, RR, TV, pressure support, Pmean
* ASA classification: 1-6
* Physical disorders under CPAP with yes or no, if yes specified:

eyes, ears, nose, throat respiratory cardiovascular musculoskeletal genitourinary skin endocrine neurological psychiatric Hypothesis

Null and alternate hypothesis:

H0: There is NO change of rSO2 during CPAP therapy. H1: There is A change of rSO2 during CPAP therapy. Type-I and -II errors and power α = 0.05 Power = 0.9 Interim analysis

* Statistical methodology Randomized observational experimental single-center clinical trial.
* Sample size calculation:

Paired t-test, mean of difference: 5%, SD of difference: 10%; Effect size of 0.5; an error probability two-sided: 0.05; Power: 0.9; total sample size: 50 patients. (5% drop-out rate included).

METHODS This randomized clinical study will include 50 subjects from 18 years onwards undergoing treatment on an ICU of the Medical University of Vienna (13C1, 13C2, 13C3, 13B1, 13I1, 9D, E11 (Neurosurgical ICU), requiring intermittent CPAP therapy. Neither the applicant, nor the clinical investigator will be involved in the decision about the indication for CPAP therapy.

The study will be carried out according to the Declaration of Helsinki (1964), and good clinical practice (GCP) guidelines, and the Equator network website recommendations including current revisions. The study protocol will be submitted to the Ethics Committee of Medical University of Vienna for ethical approval. The study will be registered with clinicaltrials.gov. The participation in the clinical study will occur independently of the medical indication for the patient's stay on the ICU. Before being admitted to the study, the subject must have consented to participate, after the nature, scope and possible consequences of the procedure have been explained in a form understandable to him or her. The patient must give consent orally and in writing. The individual's consent will be confirmed with the signature of the investigator. All subject names will be kept secret in the investigators' files. Subjects will be identified by documentation and evaluation throughout the number allotted to them during the study. The participants will be informed that the entire study data will be stored and handled confidentially. A data protocol by means of a case report form will be used.

The duration of the trial is 30min. The study starts 15min before CPAP and ends when the patient's rSO2 reaches a steady state (no change in rSO2 ± 2% for 3 min, maximal 15min) under CPAP therapy. The participants are not required to participate in any follow up visits.

This study will be carried out on patients with good access to the forehead. The NIRS measurement (IBO) will be performed on the frontal cortex on both sides of the head. Emission and detection probes have to be connected after wiping the patients forehead with a soft cloth or cotton pad. During the whole investigation the SaO2, the blood pressure (continuously invasive or non invasive in 3 minute-intervals) and the ECG will be recorded. These vital signs are a part of the routine ICU monitoring. The trial will consist of two parts i.e. with or without ventilatory assistance. The order of starting the study with or without CPAP therapy will be randomized. During each part the measurements will be performed until reaching a steady state (no change in rSO2 ± 2% for 3 min) but with a maximum duration of 15min. The examination is safe, non-invasive, pain-free and can be carried out very flexibly, quickly and cost efficiently by portable equipment. Data is collected from both the right and left hemisphere.

The device system is to be used only in accordance with the approved investigational plan and the CE-Certificate, on subjects who receive CPAP therapy and have signed an informed consent form. The use of the device is limited to the approved study investigators. After each examination interval a BGA will be performed.

The reason why this study is conducted on ICU patients is the following. Patients who suffer from respiratory deficiencies and are in need of ventilatory assistance are rarely located on normal hospital wards due to the fact that the installation of a ventilatory machine with additional CPAP mode has to be performed by specialized personnel. In addition, these patients require close monitoring, which can be guaranteed in an ICU setting.

Pregnant women, as well as individuals with severe valvular or neurological diseases will not be included in the observation study.

After the indication for CPAP-therapy is verified and the in- and exclusion criteria are checked, the patients will be recruited for the study.

The study will be divided in two data collection parts, both taken in one session.

1. 15min before CPAP:

   * starting to collect data of either continuous arterial blood pressure measurement (ABP)
   * or non invasive (NIBP) until end of study
   * starting NIRS measurement on both brain hemispheres (INVOS 5100C) until procedure is completed
   * drawing an arterial our venous (according to available access) blood sample for a blood gas analysis (BGA)
2. 15min with CPAP:

   * measurements performed in point 1. (ABP/NIBP, NIRS) will be continued
   * taking of another arterial our venous (according to available line) blood sample for a BGA

The order of point 1. and 2. (without or with CPAP) will be randomized into group 1 and group 2 in the same patient.

OPERATIONAL OBJECTIVES

1. st year: Drafting of the study proposal. Aims: - Literature search and review

   * Drafting of the study proposal
   * Detailed planning of the realization of the project

   Short description: Current literature on CPAP therapy, NIRS and rSO2 will be reviewed. The exact planning of the realization of the study will begin after the positive ethics committee vote has been received. A detailed study protocol will be written after the literature review and the performance of preliminary measurements.
2. nd year: Initiation of the project

   Aims: - Performing preliminary measurements and refining study protocol
   * Execution of the study
   * Evaluating the results

   Short description: Preliminary measurements with NIRS will be performed, after which the study protocol will be refined. According to the adapted protocol, the study will be carried out on the ICUs of the MUW.
3. rd year: Finalizing the project, statistical evaluation; Data interpretation and writing of the thesis.

Aims: - Evaluation of data

* Statistical analysis
* Interpretation of the results
* Drafting a preliminary version of the thesis
* Revision of the thesis to the supervisors's comments
* Writing a research paper to publish the study results

Short Description: Following the completion of the study, all collected data will be evaluated and subjected to statistical analysis. Future follow up studies based on these results will be drafted. The applicant will be granted time to work on his research project as part of the research group "lung".

Cooperation arrangements The project will be performed at the Department of Anesthesia, General Intensive Care and Pain Management, MUW.

Outlook and further projects

Several projects focusing on effects of rSO2 alterations in other settings are possible:

* intensive care unit therapy
* general anesthesia

REFERENCES 1-23

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing CPAP in the routine clinical treatment
* women/men on following ICUs: 13C1, 13C2, 13C3, 13B1, 13I1, 9D, E11 (neurosurgery intensive care unit)
* age above 18
* patients willing to participate

Exclusion Criteria:

* pregnancy
* present neurological disorders
* present cardiac valvular disease
* patients not willing to participate
* patients with allergies to the measurement sensor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
The changes of rSO2 under CPAP therapy | 2x15min: with and without CPAP in one session (in total about 30 minutes)

SECONDARY OUTCOMES:
rSO2 trend with and without NIV | 2x15min: with and without CPAP in one session (in total about 30 minutes)
Correlation of rSO2 to other parameters (SpO2, Bloodpressure) | 2x15min: with and without CPAP in one session (in total about 30 minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Markstaller, Prof.Dr, Study Director — MUW, Department of Anaesthesia
Locations (1):
- Medical University of Vienna, Anesthesia, Vienna, Vienna, Austria